CLINICAL TRIAL: NCT06983457
Title: Comparative Effects of Therapeutics Ultrasound and Shockwave Therapy on Pain and Quality of Life in Patients With Chronic Heel Spur Pain. A Randomized Controlled Clinical Trial
Brief Title: Comparative Effects of TherapeuticU and Shockwave Therapy on Pain and QOL in Patients With Chronic Heel Spur Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/815
Record Dates: First submitted 2025-03-29; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Heel Spur
MeSH Terms: conditions — Heel Spur | interventions — Ultrasonic Therapy; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic ultrasound (Experimental)
  Interventions: Combination Product: Therapeutic ultrasound
- Shockwave Therapy (Experimental)
  Interventions: Combination Product: Shockwave Therapy

INTERVENTIONS:
Combination Product: Therapeutic ultrasound — Participants in Group A will receive therapeutic ultrasound (TUS) as the primary intervention for managing chronic heel spur pain. The TUS treatment will be administered using a frequency of 1 MHz, which is effective for targeting deeper tissues. The intensity will range from 0.8 to 2.0 W/cm², depending on patient tolerance, and will be applied in a continuous mode to maximize thermal effects. Each treatment session will last for 4 minutes, and Treatment sessions will be conducted daily Monday through Friday for a period of 2 weeks in a series of ten treatments. The TUS application will focus on the medial calcaneal tubercle and the surrounding inflamed soft tissues to reduce pain and promote tissue healing.
  Arms: Therapeutic ultrasound
Combination Product: Shockwave Therapy — Group B (Shockwave therapy) Participants in Group B will receive extracorporeal shockwave therapy to perform the shock wave treatments, an apparatus generating a shock wave in a pneumatic manner was used, i.e., BTL-5000 SWT POWER + HIGH INTENSITY LASER 12 - to perform the shock wave treatments, an apparatus generating a shock wave in a pneumatic manner was used. Before starting the procedure, each patient was informed about the principles of the shock wave action and the possibility of side effects. Each of the project participants underwent a series of 5 treatments at 7-day intervals.
  Arms: Shockwave Therapy

SUMMARY:
This research aims to compare the effectiveness of therapeutic ultrasound (TUS) and extracorporeal shockwave therapy (ESWT) in managing chronic heel spur pain and improving patients' quality of life. Chronic heel spur pain, often associated with plantar fasciitis, is a debilitating condition that affects mobility and daily activities.

DETAILED DESCRIPTION:
The study will be conducted at Sehat Medical Complex, Lahore, over 10 months, enrolling 60 participants diagnosed with chronic heel spur pain. They will be randomly assigned into two groups: one receiving therapeutic ultrasound (10 sessions over two weeks with a frequency of 1 MHz and intensity between 0.8-2.0 W/cm²) and the other undergoing shockwave therapy (five weekly sessions with 2500 shocks per session at increasing pressure levels from 2.5 to 3.5 bars). The effectiveness of these interventions will be evaluated using the Visual Analog Scale (VAS) for pain intensity, the Foot Function Index (FFI) for functional assessment, and for quality of life. Follow-up assessments will be conducted at baseline, after the intervention (week 4), and at week 8 to evaluate both short-term and sustained treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic heel spur pain, confirmed through imaging studies (e.g., X-ray, ultrasound).
* Age range: 30-60 years. Both male and female included
* Chronic heel pain persisting for more than 1 month.
* Individuals with no prior surgical intervention for heel pain.
* Ability to provide informed consent and comply with the treatment protocol.

Exclusion Criteria:

* Presence of systemic inflammatory conditions such as rheumatoid arthritis or gout.
* History of previous steroid injection less than 6 weeks.
* prior NSAID treatment less than 1 week,
* Individuals with contraindications to ultrasound or shockwave therapy, such as pacemakers or implanted devices.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 12 Months
  A Visual Analogue Scale (VAS) is one of the pain rating scales. Pain intensity can be categorized based on VAS scores, with mild pain typically ranging from 1-3, moderate pain from 4-6, and severe pain from 7-10. Validity is 0.95% and reliability is 0.88%.
  Foot Function Index (FFI):
  A Foot Function Index (FFI) is to measure the impact of foot pathology on function in terms of pain, disability and activity restriction. The FFI is a self-administered index consisting of 23 items divided into 3 sub-scales. Validity is 0.90% and reliability is 0.85%.
Quality Of Life | 12 Months
  The 36-Item Short Form Survey (SF-36) is an outcome measure instrument that is often used, well-researched, self-reported measure of health. Each scale is directly transformed into a 0-100 scale. The higher the score the less disability i.e. a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Sehat Medical Complex, Hanjarwal campus, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No